CLINICAL TRIAL: NCT01408277
Title: A Comparison of Collagenase Santyl® Ointment Used Adjunctively to Sharp Surgical Debridement and Sharp Surgical Debridement in the Care of Diabetic Foot Wounds
Brief Title: Using Santyl on Diabetic Foot Ulcers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Healthpoint (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 017-101-09-030
Record Dates: First submitted 2011-08-02; First posted 2011-08-03 (Estimated); Results first posted 2014-05-05 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-06

CONDITIONS: Diabetic Foot Ulcers; Diabetic Foot Wounds
Keywords: Diabetic Foot Ulcers; Diabetic Foot Wounds
MeSH Terms: conditions — Diabetic Foot | interventions — Collagenases; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Santyl (Active Comparator): 2mm Santyl applied once daily.
  Interventions: Biological: Santyl
- Control (Active Comparator): Standard Care
  Interventions: Procedure: Control

INTERVENTIONS:
Biological: Santyl — 2 mm Santyl applied once daily
  Arms: Santyl
Procedure: Control — Standard Care
  Other Names: Standard Care
  Arms: Control

SUMMARY:
Subjects enrolled in this study will either use Santyl daily or follow standard care procedures for up to 6 weeks for their diabetic foot wound. After 6 weeks of treatment, the subjects will continue into the follow-up phase for an additional 6 weeks. Study doctors will look at the wound in the office each week (up to 12 weeks) to see if the wound is healing. Depending on a number of factors at each office visit, the study doctors may also use a procedure called sharp debridement to remove dead skin from the wound.

This study will test the hypothesis that daily treatment of diabetic foot wounds with Santyl will result in more rapid healing, healthier wounds, and fewer required sharp debridements over the study period than for diabetic foot wounds treated in other ways.

ELIGIBILITY:
INCLUSION CRITERIA

* Provide written informed consent, which will consist of reading, signing, and dating the informed consent document after the Investigator, sub-Investigator or other designated study staff member has explained the study procedures, risks, and contact information.
* Subjects 18 years of age or older. Subjects may be of either sex and of any race or skin type provided that their skin color, in the opinion of the Investigator, will not interfere with the study assessments.
* A target ulcer which is 0.5 cm2 - 10 cm2 inclusive (as measured at the Screening Visit) with a duration ≥ 30 days (documented in the patient's history or by patient report of onset) which requires sharp surgical debridement.
* Adequate arterial blood flow as evidenced by an ankle brachial index (ABI) of > 0.7 and ≤ 1.1. If the ABI is greater than 1.1, then a toe pressure of > 40 mmHg OR a TcPO2 ≥ 40 mmHg must be present. Either toe pressure or TcPO2 is also acceptable as a stand-alone measurement, but if both are obtained, each must meet its respective cutoff.
* Alternatively, a Doppler waveform consistent with adequate flow to the region of the foot with the target ulcer (biphasic or triphasic waveforms) is acceptable.
* A target ulcer that is not infected based on clinical assessment.
* Willing and able to make all required study visits.
* Able to follow instructions and perform the dressing changes at home or have a caregiver who can perform the dressing changes according to the protocol.
* Willing to use an appropriate off-loading device whenever necessary to keep weight off of any foot ulcers.
* History of diabetes mellitus (Type 1 or 2) requiring insulin or oral hypoglycemic medications to control blood glucose levels.
* CBC and blood chemistry values as follows:

  * Serum albumin ≥ 2.0 g/dL
  * Pre-albumin levels of ≥ 15 mg/dL
  * Alkaline phosphatase ≤ 500 U/L
  * Alanine aminotransferase (ALT) ≤ 200 U/L
  * Aspartate aminotransferase (AST) ≤ 175 U/L
  * Serum total bilirubin ≤ 3.0 mg/dL
  * Serum BUN < 75 mg/dL
  * Serum creatinine ≤ 4.5 mg/dL
  * HbA1c ≤ 12%
  * Hemoglobin (Hgb) > 8.0 g/dL
  * WBC > 2.0 x 109/L
  * Absolute neutrophil count > 1.0 x 109/L
  * Platelet count > 50 x 109/L

EXCLUSION CRITERIA

* Contraindications or hypersensitivity to the use of the study medications or their components.
* Target ulcer does not require debridement.
* Uncontrolled bleeding disorder.
* Cellulitis of the target wound, lymphangitic streaking, deep tissue abscess, gangrene, or infection of muscle, tendon, joint or bone.
* Infection with systemic toxicity or metabolic instability (e.g., fever, chills, tachycardia, hypotension, confusion, vomiting, leukocytosis, acidosis, severe hyperglycemia, azotemia).
* Any of the following:

  * Target ulcer tunneling
  * Target ulcer requires hyperbaric or negative pressure therapy per the investigator's medical judgment
  * Target ulcer is on the heel and cannot be offloaded
  * Target ulcer is over a Charcot deformity which cannot be offloaded
* NOTE: A heel ulcer or an ulcer over a Charcot is not excluded unless effective offloading is not possible.
* Current, ongoing osteomyelitis of the target foot as determined by medical history.
* Participation in another investigational clinical study within thirty (30) days of the Screening Visit.
* A target ulcer which involves underlying tissues (i.e., fat, fascia, tendon, muscle, bone).
* A target ulcer on a non-neuropathic foot (neuropathic defined as inability to perceive 10 grams pressure using a Semmes-Weinstein 5.07 or equivalent monofilament in the periwound area).
* NOTE: Monofilament test result must be documented.
* Diagnosis of chronic granulomatous disease, leukocyte adhesion defects, or severe neutropenia.
* Current treatment (at the time of the Screening Visit) with any of the following:

  * Systemic corticosteroids
  * Immunosuppressive agents
  * Chemotherapeutic agents
  * Antiviral agents
  * Platelet-derived growth factor (e.g., Regranex)
  * Living skin equivalent (e.g., Apligraf)
  * Dermal substitute (e.g., Dermagraft, Integra, etc.)
  * Systemic antibiotic therapy or topical antibiotic treatment of the target ulcer
* Radiation therapy to the target lower extremity within 30 days prior to screening The Medical Monitor and/or Investigator may declare any subject ineligible for a valid medical reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2011-08; Primary Completion 2012-11 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert B Slade, MD, Study Chair — Healthpoint
Locations (7):
- United States (7):
  - Associated Foot and Ankle Specialists, Phoenix, Arizona
  - Aung Foothealth Clinics, Tucson, Arizona
  - Foot Healthcare Associates, PC, Southfield, Michigan
  - Overlook Hospital Wound Care Center, Summit, New Jersey
  - UNTHSC Fort Worth, Fort Worth, Texas
  - Robert Wunderlich, San Antonio, Texas
  - Endeavor Clinical Trials, San Antonio, Texas

REFERENCES:
- [Derived] Motley TA, Gilligan AM, Lange DL, Waycaster CR, Dickerson JE Jr. Cost-effectiveness of clostridial collagenase ointment on wound closure in patients with diabetic foot ulcers: economic analysis of results from a multicenter, randomized, open-label trial. J Foot Ankle Res. 2015 Feb 28;8:7. doi: 10.1186/s13047-015-0065-x. eCollection 2015. PMID 25767565

RESULTS

PARTICIPANT FLOW:
Groups:
- Santyl: Collagenase (SANTYL®) Ointment
Period: Overall Study
Arm/Group | Santyl | Control
Started | 28 | 27
Completed | 20 | 23
Not Completed | 8 | 4
Not completed — Adverse Event | 3 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Protocol Violation | 2 | 0

BASELINE CHARACTERISTICS:
Population: 20 subjects from each group was a priori considered to be a number sufficient to detect an effect size (Cohen's d) of 0.80, regarded as a large effect, with α = 0.05 and 1-β = 80%.
Groups:
- Total: Total of all reporting groups
Arm/Group | Santyl | Control | Total
Number analyzed (Participants) | 28 | 27 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 20 | 42
  >=65 years | 6 | 7 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 21 | 20 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 9
  Not Hispanic or Latino | 23 | 23 | 46
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 25 | 22 | 47
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 28 | 27 | 55

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change in Wound Area
Description: Wound area was measured using the ARANZ Silhouette digital wound imaging and measurement device. The average percent (%) of change from baseline of the target wound area at the end of the 6-week treatment period and the end of the entire 12-week study period respectively, was calculated using a two-way ANCOVA model.
Time Frame: 6 and 12 weeks
Population: Primary analysis was based on the Intent-to-treat dataset which consisted of all subjects randomized to treatment.
Measure: Mean (Standard Error); unit: percentage of change in wound area
Groups:
- Santyl®: Collagenase (Santyl®) Ointment
- Control: Control = Standard Care
  Standard Care is defined as the standard wound care protocol for chronic wounds used by each Investigator, in their clinic (e.g., wet-to-dry, compression, sharp debridement, etc.).
Arm/Group | Santyl® | Control
Number analyzed (Participants) | 28 | 27
percentage of change in wound area
  % change at end of 6 weeks | -68 (6.3) | -36 (20.4)
  % change at end of 12 weeks | -61 (9.6) | -46 (18.3)

ADVERSE EVENTS:
Time Frame: 12 weeks
Groups:
- Santyl: Collagense (Santyl®) Ointment
Arm/Group | Santyl | Control
Serious Adverse Events (participants affected / at risk) | 3/28 | 4/27
Other Adverse Events (participants affected / at risk) | 7/28 | 6/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Santyl (N=28) | Control (N=27)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Gangrene (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Santyl (N=28) | Control (N=27)
Cellulitis (Infections and infestations) | 2 (2) | 2 (2)
Osteomyelitis (Infections and infestations) | 1 (1) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Wound complication (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No